CLINICAL TRIAL: NCT06671353
Title: Randomized, Controlled Trial of a Video Decision Support for Advance Care Planning in Geriatric Patients With Frailty
Brief Title: Video Decision Support for Advance Care Planning in Geriatric Patients With Frailty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202312031RIND
Record Dates: First submitted 2024-10-28; First posted 2024-11-04 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Frail Elderly
Keywords: frailty; advance care planning; shared decision making
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- with video decision aid (Active Comparator): video decision aid
  Interventions: Behavioral: video decision aid

INTERVENTIONS:
Behavioral: video decision aid — video decision aid for advance care planning
  Arms: with video decision aid

SUMMARY:
As the proportion of the aging population continues to rise, age-related frailty syndrome, characterized by a decline in the function of multiple physiological systems and accompanied by vulnerability to stress, has become a significant issue. It has been associated with higher mortality rates, hospitalization rates, risk of falls, occurrence of fractures, decreased mobility, depression, cognitive decline, dementia, loneliness, and admission to long-term care facilities. Advance care planning is a thoughtful and communicative process that helps individuals, while still cognitively capable, to pre-determine and express their preferences for medical care in the event of future incapacity. With the ongoing development in the field of frailty and the rapid aging of the population, the increasing age may be accompanied by severe illnesses, symptom burden, functional dependence, caregiver burden, and extensive medical utilization. The importance of advance care planning is increasingly emphasized, but its implementation and promotion remain challenging. In addition to systematic promotion from a policy perspective, tools to assist patients in decision-making have been proposed. Video decision aids can encourage people to engage in advance care planning by sparking conversations about informed consent and helping individuals contemplate the choices they may face. Video decision aids can also assist individuals in envisioning future scenarios and reflecting on their decisions. Previous randomized controlled trials have explored the benefits of such video tools for specific patient populations, such as cancer patients, heart failure patients, and elderly individuals hospitalized. However, there is a need for innovative approaches to enhance the knowledge, willingness, and actual signing rates of advance care planning for frail elderly individuals. This study aims to develop a video decision aid specifically tailored for the elderly frail population undergoing advance care planning.

Through a randomized controlled trial, the study aims to validate its actual benefits, expecting to assist the elderly frail population in understanding and expressing their willingness for advance care planning, increasing the actual willingness to sign advance directives, and helping clinical healthcare teams achieve person-centered, high-quality care for this population.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 65 y/o can communicate and sign informed consent diagnosed to be frailty with clinical frailty scale 4-7

Exclusion Criteria:

* impaired visual acuity or hearing that can't watch video had signed advance decision before

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients completed advance decision | from enrollment to 4 weeks after watching video decision aid
  The advance decision must be completed by the patients and uploaded to the National Health insurance system

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Research Ethics Committee, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
the data will include personal data

REFERENCES:
- [Background] Thompson JS, Matlock DD, McIlvennan CK, Jenkins AR, Allen LA. Development of a Decision Aid for Patients With Advanced Heart Failure Considering a Destination Therapy Left Ventricular Assist Device. JACC Heart Fail. 2015 Dec;3(12):965-76. doi: 10.1016/j.jchf.2015.09.007. PMID 26671675